CLINICAL TRIAL: NCT03179488
Title: Intensity Matters: Therapist-dependent Dose of Spinal Transcutaneous Electrical Nerve Stimulation
Brief Title: Therapist-dependent Dose of Spinal TENS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Castilla-La Mancha (Other)
Collaborators: Hospital Nacional de Parapléjicos de Toledo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: ddsm22
Record Dates: First submitted 2017-06-05; First posted 2017-06-07 (Actual); Last update posted 2017-07-05 (Actual); Status verified 2017-06

CONDITIONS: Transcutaneous Electrical Nerve Stimulation; Spinal Cord Stimulation; Dose-response Relationship

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled, crossover trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spinal TENS stimulation (Experimental): Spinal TENS stimulation: A constant voltage and a symmetric biphasic current of 200 microseg pulse-width at a frequency of 100Hz. The intensity will increase until participants report a "strong but comfortable" sensation, just below motor threshold.
  Interventions: Device: Spinal TENS
- Sham stimulation (Sham Comparator): The same procedures as experimental group, but but will be applied a sham electrical stimulation increasing the current intensity until sensory perception of the stimulus, and then decreased to zero where it will fix until the end of the stimulation.
  Interventions: Device: Sham stimulation

INTERVENTIONS:
Device: Spinal TENS — Spinal TENS stimulation over back through the electrotherapy device Myomed 932. (Enraf-Nonius, Delft, Netherlands)
  Arms: Spinal TENS stimulation
Device: Sham stimulation — Sham stimulation over back through the electrotherapy device Myomed 932. (Enraf-Nonius, Delft, Netherlands)
  Arms: Sham stimulation

SUMMARY:
The intensity used during transcutaneous electrical nerve stimulation (TENS) in both, clinical practice and research studies, is often based on subjective commands such as "strong but comfortable sensation". There is not consensus regarding the effectiveness dose of TENS

DETAILED DESCRIPTION:
Twenty healthy volunteers will divide into two groups: Therapist 1 and Therapist 2. Both therapist will apply spinal TENS and sham stimulation for 40min in random order to each subject, at an intensity to produce a "strong but comfortable sensation".

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers between 18 and 60 years old

Exclusion Criteria:

* Musculoskeletal pathology of the lower limbs
* History of neuromuscular disease
* Unable to tolerate electrical current
* Allergy to the electrode material
* Pacemaker or any implanted device
* Epilepsy
* Neurotrauma
* Recent surgical procedures
* Pain affecting the lower limbs or lower back
* Diabetes
* Pregnancy
* Cancer

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-07-03 (Actual); Primary Completion 2017-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Baseline Current Density | At the onset (0min) of the Spinal TENS session
  Current density (mA/cm2) is obtained by a mathematical operation which reflects the applied current intensity divided by the electrode area (45cm2)
Final Current Density | At the end (40min) of the Spinal TENS session
  Current density (mA/cm2) is obtained by a mathematical operation which reflects the applied current intensity divided by the electrode area (45cm2)

SECONDARY OUTCOMES:
Baseline Maximal peak-to-peak soleus H-reflex | baseline at 0min
  H-reflex data are obtained by electromyography activity (EMG). The EMG electrode is fixed on triceps surae. The stimulator electrode is fixed on the peroneus nerve, in the popliteal fossa.
Baseline Maximal peak-to-peak soleus M wave | baseline at 0min
  M wave ddata are obtained by electromyography activity (EMG). The EMG electrode is fixed on triceps surae. The stimulator electrode is fixed on the peroneus nerve, in the popliteal fossa.
Baseline Normalized H-reflex response | baseline at 0min
  Normalized H-reflex response data are obtained by electromyography activity (EMG). The EMG electrode is fixed on triceps surae. The stimulator electrode is fixed on the peroneus nerve, in the popliteal fossa.
During Maximal peak-to-peak soleus H-reflex | during treatment at 33min
  H-reflex data are obtained by electromyography activity (EMG). The EMG electrode is fixed on triceps surae. The stimulator electrode is fixed on the peroneus nerve, in the popliteal fossa.
During Maximal peak-to-peak soleus M wave | during treatment at 33min
  M wave data are obtained by electromyography activity (EMG). The EMG electrode is fixed on triceps surae. The stimulator electrode is fixed on the peroneus nerve, in the popliteal fossa.
During Normalized H-reflex response | during treatment at 33min
  Normalized H-reflex response data are obtained by electromyography activity (EMG). The EMG electrode is fixed on triceps surae. The stimulator electrode is fixed on the peroneus nerve, in the popliteal fossa.
Post-treatment Maximal peak-to-peak soleus H-reflex | Immediately after treatment at 40 min
  H-reflex data are obtained by electromyography activity (EMG). The EMG electrode is fixed on triceps surae. The stimulator electrode is fixed on the peroneus nerve, in the popliteal fossa.
Post-treatment Maximal peak-to-peak soleus M wave | Immediately after treatment at 40 min
  M wave data are obtained by electromyography activity (EMG). The EMG electrode is fixed on triceps surae. The stimulator electrode is fixed on the peroneus nerve, in the popliteal fossa.
Post-treatment Normalized H-reflex responseMaximal peak-to-peak soleus H-reflex | Immediately after treatment at 40 min
  Normalized H-reflex response data are obtained by electromyography activity (EMG). The EMG electrode is fixed on triceps surae. The stimulator electrode is fixed on the peroneus nerve, in the popliteal fossa.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Avendaño-Coy, PhD, Study Director — University of Castilla-La Mancha; Diego Serrano-Muñoz, MsC, Principal Investigator — Hospital Nacional de Parapléjicos de Toledo
Locations (1):
- Juan Avendaño-Coy, Toledo, Spain

IPD SHARING:
Plan to Share IPD: No